CLINICAL TRIAL: NCT06642701
Title: Electrical Impedance Imaging Techniques in Guiding the Use of Chest Physiotherapy in Patients with Pneumonia: a Randomized Controlled Study
Brief Title: Electrical Impedance Imaging Techniques in Guiding the Use of Chest Physiotherapy in Patients with Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jingyi Ge, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-2-2252
Record Dates: First submitted 2024-08-20; First posted 2024-10-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EIT-guided group (Experimental): Physical therapy guided by EIT
  Interventions: Device: Electrical Impedance Tomography; Behavioral: chest physiotherapy
- Non-EIT-guided group (Other): Traditional physical therapy
  Interventions: Behavioral: chest physiotherapy

INTERVENTIONS:
Device: Electrical Impedance Tomography — According to the results of traditional assessment, physiotherapists and clinicians discussed the EIT results to give respiratory rehabilitation chest physiotherapy
  Arms: EIT-guided group
Behavioral: chest physiotherapy — Conventional assessment by physical therapists was followed by respiratory rehabilitation chest physiotherapy.Chest physical therapy for respiratory rehabilitation includes postural drainage, cough technique, forced expiratory technique, positive expiratory pressure, high-frequency chest wall compression, chest tapping, vibration, active breathing cycle technique, etc. All chest physiotherapy was performed by 1 therapist.

SUMMARY:
In this study, electrical impedance tomography (EIT), a noninvasive and nonradiative technology, is applied to guide the accurate respiratory rehabilitation of pneumonia. On the basis of traditional physical assessment, physiotherapists introduce EIT as an auxiliary imaging technology into the field of rehabilitation, which can increase the accurate understanding of ventilation conditions of local lung lesions, so as to optimize physical therapy methods, which is conducive to the improvement of patients' symptoms, the improvement of lesions, and the improvement of patients' quality of life.

DETAILED DESCRIPTION:
According to the results of traditional assessment, physiotherapists and clinicians discussed the EIT results to give respiratory rehabilitation chest physiotherapy, and adjusted the treatment according to the results of T2 and T3 review. EIT has dynamic monitoring charts and communicates with patients about the changes after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Meet the diagnostic criteria of CAP：(1) community onset; (2) pneumonia-related clinical manifestations: recent onset of cough, expectoration or worsening of symptoms of preexisting respiratory diseases, with or without sputum purulence, chest pain, dyspnea or hemoptysis; Fever; Signs of lung consolidation and/or moist rales were heard; Peripheral white blood cell count > 10×109/L or < 4×109/L, with or without nuclear shift to the left. (3) Chest imaging examination: new patchy infiltrates, lobar/segmental consolidation, ground glass opacity or interstitial changes, with or without pleural effusion. The clinical diagnosis was established when any one of (1), (3) or (2) was met, excluding pulmonary tuberculosis, lung tumor, non-infectious interstitial lung disease, pulmonary edema, atelectasis, pulmonary embolism, pulmonary eosinophil infiltration and pulmonary vasculitis.
* Meet the diagnostic criteria of HAP： Referring to the Chinese adult (2018 edition), it refers to the new-onset pneumonia within 48 hours after admission of patients who have not received invasive mechanical ventilation during hospitalization and are not in the incubation period of pathogenic infection. "That is, new or progressive infiltrates appear in the lung, and there are more than two of the following symptoms: fever, increased neutrophils (>10×109/L) or decreased neutrophils (<5×109/L), purulent sputum.
* The need for chest physical therapy for patients with pneumonia was determined jointly by the rehabilitation treatment team including clinicians, rehabilitation physicians and therapists, and the consent of patients and their families was obtained.

Exclusion Criteria

* Invasive or noninvasive mechanical ventilation；
* Ventilator-associated pneumonia；
* permanent or temporary cardiac pacemaker installed in the body；
* Moderate or massive pleural effusion；
* Severe pneumonia: disturbance of consciousness; Respiratory rate ≥ 30 breaths /min; PaO2<60 mmHg, PaO2/FiO2<300, need mechanical ventilation treatment; Systolic arterial pressure <90 mmHg; Complicated with septic shock; Chest X-ray showed bilateral or multi-lobar involvement or lesion enlargement ≥ 50% within 48 hours after admission；Urine output<20 mL/h, or <80 mL/4 h, or complicated with acute renal failure requiring dialysis treatment；Patients with one or more of these parameters were diagnosed as severe disease；
* body mass index> 30kg/m2；
* Lung cancer；
* Acute exacerbation of chronic obstructive pulmonary disease and acute exacerbation of bronchial asthma；
* Viral pneumonia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Clinical pulmonary infection score | Before respiratory rehabilitation chest physiotherapy (T1), on days 3 (T2) and 7 (T3) after the start of treatment.
  CPIS is a comprehensive assessment of the severity of infection based on clinical, radiological, and microbiological criteria, including body temperature, white blood cell count, tracheal secretions, oxygenation, chest X-ray, progression of pulmonary infiltrates, and tracheal aspirate culture. The maximum score was 12 and the minimum score is 0 points.. It is of great significance in the diagnosis, treatment and evaluation of pneumonia, and has high application value.The higher the CPIS score, the more serious the patient's clinical condition is and the more timely treatment is needed. When the CPIS score is ≤6, the discontinuation of antibiotics can be considered.

OTHER OUTCOMES:
Length of stay | From admission to discharge, assessed up to 1 day
  The length of stay for each patient.
Short Form 36 | At baseline and at week 2.
  The Short Form-36 (SF-36) scale was used to assess quality of life. The lowest score represents the worst health status. SF-36 measurement was performed twice, before and after treatment.
Satisfaction with treatment | Evaluation was conducted 12 hours before discharge.
  Using the Australian respiratory rehabilitation package, divided into 5 items, each item 5 points, a total of 25. The original questionnaire contained six items on which patients rated their satisfaction with respiratory rehabilitation on a scale of 1 strongly disagree to 5 strongly agree.
Regional Ventilation distribution | From baseline measurements to immediately after the end of treatment (15 minutes)
  Difference in regional ventilation distribution before and after institution of physical therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jingyi Ge, Principal Investigator — Beijing Rehabilitation Hospital of Capital Medical University
Locations (1):
- Jingyi Ge, Beijing, China

IPD SHARING:
Plan to Share IPD: No